CLINICAL TRIAL: NCT02764385
Title: Using a Teachable Moment Communication Process to Improve Outcomes of Quitline Referrals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Susan Flocke, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RES206807
Record Dates: First submitted 2016-04-14; First posted 2016-05-06 (Estimated); Results first posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Smoking; Tobacco Dependence
MeSH Terms: conditions — Smoking; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AAC only (Other): This is a system-based intervention that involves changes in the EHR regarding documenting tobacco assessment and the capability to order an eReferral to the Quitline. This system-based intervention also changes the role of the medical technical assistant.
  Interventions: Other: AAC
- AAC + TMCP (Other): The Teachable Moment Communication Process is a clinician-focused intervention designed to guide an approach to discussing smoking cessation during routine primary care visits.
  Interventions: Other: Teachable Moment Communication Process; Other: AAC

INTERVENTIONS:
Other: Teachable Moment Communication Process — A clinician-focused intervention designed to guide an approach to discussing smoking cessation during routine primary care visits.
  Arms: AAC + TMCP
Other: AAC — A system-based change to the EHR that allows for eReferral to the Quitline coupled with role and process changes for medical technical assistants

SUMMARY:
This study will compare the effectiveness of two approaches for delivering smoking cessation advice in the primary care setting. Ask-Advise-Connect (AAC) is a strategy that uses the electronic health record (EHR) to prompt clinical staff to Ask if the patient smokes, Advise them to quit and, if they're interested, Connect them to Quitline (QL) counseling services. The connection occurs when a QL counselor is notified of the patient's interest, and then calls the patient to enroll in treatment. AAC has been shown to be very effective at enrolling patients, however, it was found that less than 42% of patients who agreed to be referred were successfully contacted by the QL after 5 call attempts. This indicates that many patients that are referred are not ready for cessation, but may feel obligated to accept the referral from their primary care team. This presents an opportunity to improve the patient centeredness of the referral process.

To overcome these limitations, the investigators propose pairing it with a patient-centered smoking cessation approach called the Teachable Moments Communication Process (TMCP). The investigators' team developed this communication strategy, which incorporates patients' concerns into a partnership-oriented discussion about smoking cessation. The investigators propose that combining these two approaches could increase appropriate referrals to the QL, increase the likelihood of successful patient contact and enrollment, and increase the patient's rating of the value of the experience.

DETAILED DESCRIPTION:
The investigators specifically aim to:

1. Improve delivery and documentation of smoking cessation advice and assistance to socially and economically disadvantaged patients using an AAC approach integrated into the EHR.
2. Test the effect of combining the TMCP with AAC on process, Quitline referral and smoking outcomes.
3. Examine the narratives of subgroups of individuals to better understand the referral experience and identify ways to improve it.

The investigative research team will conduct a randomized trial to implement these strategies with 8 clinics serving more than 25,000 patients who smoke. The investigators first implement the AAC system change intervention and then use a stepped wedge design to implement the TMCP in 8 clinics that are randomly assigned to a time point (step) for receiving the TMCP intervention. The investigators will collect data via patient survey, EHR and Quitline. The investigators also will conduct in-depth interviews with sub-groups of patients to inform ways to improve the referral process. With mounting demand for systems-based solutions for providing tobacco cessation assistance, it is urgent to understand how to use a systems approach like the AAC in a way that attends to the patient experience. The findings from this study will be useful to clinicians, patients, healthcare systems, and health insurance plans.

ELIGIBILITY:
Inclusion Criteria:

* All adults age 18+ who present for visits at participating clinics

Exclusion Criteria:

* Any individual under 18 years of age presenting for a clinic visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15786 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Flocke, PhD, Principal Investigator — Oregon Health and Science University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flocke SA, Albert EL, Lewis SA, Love TE, Rose JC, Kaelber DC, Seeholzer EL. A cluster randomized trial evaluating a teachable moment communication process for tobacco cessation support. BMC Fam Pract. 2021 May 4;22(1):85. doi: 10.1186/s12875-021-01423-x. PMID 33947346

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AAC Only | AAC + TMCP
Started | 9145 | 6641
Completed | 9145 | 6641
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AAC Only | AAC + TMCP | Total
Number analyzed (Participants) | 9145 | 6641 | 15786
Age, Customized [Count of Participants; unit: Participants]
  18-34 years | 1697 | 1123 | 2820
  35-64 years | 6532 | 4675 | 11207
  65+ years | 916 | 843 | 1759
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5300 | 3885 | 9185
  Male | 3845 | 2756 | 6601
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4194 | 3177 | 7371
  White | 4334 | 2993 | 7327
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 617 | 471 | 1088

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Contacted for Quitline Enrollment
Description: The number of patients contacted by the Quitline among those ready to quit and who accepted a referral to the quitline
Time Frame: Every visit until end of study, up to 6 months post TMCP implementation
Population: unit is the patient; among referrals received by the quitline, documented as contacted.
Measure: Count of Participants; unit: Participants
Arm/Group | AAC Only | AAC + TMCP
Number analyzed (Participants) | 1393 | 426
Participants | 273 | 59
Statistical Analysis 1: Comparison: AAC Only vs AAC + TMCP; Test type: Superiority; Odds Ratio (OR) = 1.87, 95% CI 2-sided [1.73 to 2.01]
Statistical Analysis 2: Comparison: AAC Only vs AAC + TMCP; Test type: Superiority; p = .05, Regression, Logistic; We adjust for clustering of visit within clinician and clinical site and the stepped wedge study design using generalized estimating equation methods; Odds Ratio (OR) = .68, 95% CI 2-sided [.45 to 1.02]

2. Secondary Outcome: Number of Patients With Documentation of Brief Advice
Description: The number of patients that use tobacco with documentation of brief advice
Time Frame: Every visit until end of study, up to 6 months post TMCP implementation
Population: number of smokers
Measure: Count of Participants; unit: Participants
Arm/Group | AAC Only | AAC + TMCP
Number analyzed (Participants) | 9145 | 6641
Participants | 7086 | 5579
Statistical Analysis 1: Comparison: AAC Only vs AAC + TMCP; Test type: Superiority; Odds Ratio (OR) = 1.87, 95% CI 2-sided [1.73 to 2.10]

ADVERSE EVENTS:
Description: All cause mortality, serious and other adverse events were not monitored.
Arm/Group | AAC Only | AAC + TMCP
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Intent to treat analyses are presented. Of the 60 eligible clinicians, 44 had exposure to the Teachable Moment Communication Process training. Uptake and use of the communication process during patient visits was limited (less than 10% of eligible visits). This makes it difficult to evaluate the added value of the Teachable Moment Communication Process intervention over and above the Ask-Advise-Connect approach.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/85/NCT02764385/Prot_SAP_000.pdf